CLINICAL TRIAL: NCT04015570
Title: A Randomized Controlled Trial to Study the Efficacy and Safety of Plasma Exchange Compared to Standard Medical Therapy in Patients With Severe Drug Induced Liver Injury With or Without Underlying Chronic Liver Disease.
Brief Title: Efficacy and Safety of Plasma Exchange Compared to Standard Medical Therapy in Patients With Severe Drug Induced Liver Injury With or Without Underlying Chronic Liver Disease.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ILBS-Cirrhosis-24
Record Dates: First submitted 2019-07-08; First posted 2019-07-11 (Actual); Last update posted 2019-07-11 (Actual); Status verified 2019-07

CONDITIONS: Chronic Liver Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High Volume Plasma Exchange with SMT (Experimental): PLASMA EXCHANGE is therapeutic procedure in which blood of the patient is passed through a medical device which separates plasma from other components of blood. The plasma is removed and replaced with a replacement solution such as colloid solution (e.g., albumin and/or plasma) or a combination of crystalloid/colloid solution.Plasma exchange leads to removal of abnormal circulating plasma factor or a physiologic factor produced in excess (IG, NH3,protein bond toxins )and also exert a immunomodulatory activity.
  Standard Medical Treatment (Albumin + High Caloric Diet)
  Interventions: Biological: High Volume Plasma Exchange; Other: Standard Medical Treatment
- Standard Medical Treatment (Active Comparator): Standard Medical Treatment (Albumin + High Caloric Diet)
  Interventions: Other: Standard Medical Treatment

INTERVENTIONS:
Biological: High Volume Plasma Exchange — PLASMA EXCHANGE is therapeutic procedure in which blood of the patient is passed through a medical device which separates plasma from other components of blood. The plasma is removed and replaced with a replacement solution such as colloid solution (e.g., albumin and/or plasma) or a combination of crystalloid/colloid solution.Plasma exchange leads to removal of abnormal circulating plasma factor or a physiologic factor produced in excess (IG, NH3,protein bond toxins )and also exert a immunomodulatory activity
  Arms: High Volume Plasma Exchange with SMT
Other: Standard Medical Treatment — Standard Medical Treatment (Albumin+High caloric diet)

SUMMARY:
In this randomized study subject will be randomized into two groups Group A will receive Standard Medical Treatment (Albumin + High Caloric Diet) Group B will continue Standard Medical Treatment with High Volume Plasma Exchange. All other interventions will be at the discretion of clinicians.

ELIGIBILITY:
Inclusion Criteria:

* Age-18-70 years
* Preferably Biopsy proven or history suggestive of DILI (Drug Induced Liver Injury)

  1. Grade IV DILI With T.B > 15
  2. DILI Manifesting as ACLF (Acute on chronic Liver failure) /ALF (Acute Liver Failure) with no transplant option

Exclusion Criteria:

* Evidence of active infection
* Refusal of consent or assent
* Patients with clinical suspicion of irreversible brain injury
* Pregnancy
* HCC (Hepatocellular Carcinoma) or any other malignancy
* Kidney failure
* Portal vein thrombosis
* Upper GastroIntestinal bleed
* Transplant

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-07-09 (Actual); Primary Completion 2020-07-01 (Estimated); Study Completion 2020-07-01 (Estimated)

PRIMARY OUTCOMES:
Transplant free survival in both group | Day 28

SECONDARY OUTCOMES:
Number of participants with the development of organ dysfunction or failure in both group | Day 7
Number of participants with the development of organ dysfunction or failure in both group | Day 15
Number of participants with the development of organ dysfunction or failure in both group | Day 28

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Liver & Biliary Sciences, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: Undecided